CLINICAL TRIAL: NCT00449319
Title: AML Treatment in Untreated Adult Patients According to EORTC-GIMEMA Protocols AML8 and AML10
Brief Title: AML Treatment in Untreated Adult Patients
Acronym: LAM99P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LAM99P
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Leukemia, Myelocytic, Acute
Keywords: AML; adult; Hydroxyurea; Transplant; Toevaluate biological characteristics at diagnosis.; To identify genetic alterations with prognostic relevance.; To follow up cases monitoring minimal disease during remission.; To evaluate pretreatment therapy in terms of response rate and toxicity.; Disease free survival.; Overal survival.
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Daunorubicin; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Identification of appropriate therapies according to risks factors
Drug: Daunorubicine
Procedure: Transplant

SUMMARY:
The present therapy intends to be an homogeneous treatment for AML patients based on a pretreatment with hydroxiurea plus an induction therapy with the standard arm with Daunorubicine as according to EORTC-GIMEMA AML10 study.

The post-remissional treatment is based on transplant with HLA compatible donor is foreseen for all patients and autologous transplant for those without HLA compatible donor available.

DETAILED DESCRIPTION:
GIMEMA treatment for adult (15-60 yrs) AML patients included a 3-drug induction cycle with DNR (50 mg/m2 d 1, 3, 5), cytarabine (100 mg/m2 d1-10), etoposide (100 mg/m2 d1-5) followed by an intensive consolidation with cytarabine (500 mg/m2/q12 hrs d1-d6) and the same anthracycline as in induction on d 4-6. Following consolidation, eligible pts (age <45 or 55 yrs) with a HLA compatible sibling had to be allografted, the others, had to be autografted with autologous peripheral stem cell (PSC) collected during recovery from consolidation.

BM and PB samples at diagnosis were centralized according to a national GIMEMA original study planned with the aim to accurately evaluate biological characteristics at diagnosis and to identify genetic alterations with prognostic relevance and to follow up cases monitoring minimal disease during remission. To allow the adequate collection and sending of samples before starting intensive chemotherapy, all patients received a 5-day pretreatment consisting of hydroxiurea (HU) at the dosage of 2 g/m2/day, also effective for "debulkying" of disease.

ELIGIBILITY:
Inclusion Criteria:

* AML "de novo" with bone marrow blasts <=30%
* Performance status: 0-3
* FAB subtype: all except M3
* Written informed consent

Exclusion Criteria:

* age <15 years and >= 61 years
* pretreated AML with chemiotherapy (except Idrossiurea) or radiotherapy or corticosteroids for more than 7 days.
* diagnosis of acute promyelocitic leukemia (M3)
* Performance status = 4
* Uncontrolled infection

Ages: 15 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1998-11 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Franco MANDELLI, Pr., Principal Investigator — Gruppo Italiano Malattie EMatologiche dell'Adulto
Locations (36):
- Italy (36):
  - Prof. Mozzana, Gallarate
  - Dr. De Blasio, Latina
  - Prof. Nalli, Lodi
  - Prof. Bordigon, Milan
  - Dr Miraglia, Napoli
  - Dr. Mettivier, Napoli
  - Dr.ssa Mastrullo, Napoli
  - Prof. Pane, Napoli
  - Prof. D'Arco, Nocera Inferiore
  - Dr Avanzi, Novara
  - Dr. Gabbas, Nuoro
  - Prof. Saglio, Orbassano
  - Dr Mirto, Palermo
  - Prof. Citarrella, Palermo
  - Prof. Mariani, Palermo
  - Prof. Rizzoli, Parma
  - Pr. Mecucci, Perugia
  - Prof. Falini, Perugia
  - Prof. Martelli, Perugia
  - Dr. Fioritoni, Pescara
  - Pr. Petrini, Pisa
  - Dr. Ricciuti, Potenza
  - Dr. Nobile, Reggio Calabria
  - Dr. Andriani, Roma
  - Dr. Majolino, Roma
  - Pr. Amadori, Roma
  - Pr. Annino, Roma
  - Pr. Leone, Roma
  - Pr. Lo Coco, Roma
  - Dr. Santoro, Rozzano
  - Pr. Carella, San Giovanni Rotondo
  - Pr. Longinotti, Sassari
  - Dr Epis, Sondalo
  - Dr. Russo, Taormina
  - Dr Mazza, Taranto
  - Pr. Boccadoro, Torino